CLINICAL TRIAL: NCT03710668
Title: Gut Microbiota and Parkinson's Disease
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Alaa E Ahmed (Other)
Responsible Party: Sponsor-Investigator, Alaa E Ahmed, Doctor, Assiut University
Organization: Assiut University (Other)
Other Study IDs: GMAPD
Record Dates: First submitted 2018-10-08; First posted 2018-10-18 (Actual); Last update posted 2018-10-18 (Actual); Status verified 2018-10

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Stool Sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: MRI if indicated — MRI brain if indicated

SUMMARY:
Over the past decade, experimental data has suggested a complex and bidirectional interaction between the gastrointestinal (GI) tract and the central nervous system (CNS), the so-called "Gut- Brain axis." . Changes in the gut microbiota composition may cause alterations in the gut barrier function and intestinal permeability, affecting not only GI epithelial cells and immune system, but also the ENS including both neurons and glial cells . The bidirectional brain-gut-microbiota axis interactions modulate pro- and anti-inflammatory responses. It has been suggested that the gut microbiota changes associated with intestinal inflammation may contribute to the initiation of α-syn misfolding. There is a growing number of evidence confirming that the gut microbiota alterations precede or occur during the course of PD. Importantly, some genetic risk factors may play a crucial role in the interactions between the brain-gut-microbiota axis with respect to gut inflammation. It has been also shown that the methylation status in the SNCA promoter region may affect α-syn expression and the risk for PD. Therefore, a potential role of the gut microbiota as an epigenetic factor influencing DNA methylation may be speculated. Moreover, genetic variant of the component of innate immune system - TREM2 (Triggering Receptor Expressed on Myeloid cells) has been reported to be associated with a higher risk for PD. The ε4 allele of apolipoprotein E (ApoE) has been shown to increase the risk for dementia in synucleinopathies such as PD. Potentially, ApoE genotype, by influencing bile acid secretion, could affect the composition of the gut microbiota to favor the development of organisms triggering misfolding. Moreover, three single nucleotide polymorphisms in CARD15 gene, known to be associated with Crohn's disease, have been also shown to be over-expressed in PD patients, supporting the observation that GI inflammation contributes to the pathogenesis of PD.

DETAILED DESCRIPTION:
* Normal gut microbiota is essential in preventing colonization of the harmful bacteria by competing with them for vital resources such as food and growth factors .
* Another way that gut microbiota can enhance the function of the intestinal barrier is through protecting and improving epithelial tight junctions.
* Infection and disease can also briefly affect natural gut flora composition and consequently have harmful effects on the host . Toxins produced by pathogenic microorganisms and the focal inflammation created by immune responses to them can increase gut permeability.

Impaired intestinal barrier function and consequent increased gut permeability can lead to increased translocation of gut bacteria across the intestinal wall and into the mesenteric lymphoid tissue. Furthermore, increased permeability of the gut can also increase the translocation of metabolic products such as lipopolysaccharide (LPS) or neuroactive peptides created by the bacteria that can alter the activity of the enteric nervous system (ENS) and central nervous system (CNS). Increased exposure of the ENS or mucosal immune cells to bacteria can provoke an immune response that can lead to release of inflammatory cytokines and activation of the vagus nerve and spinal afferent neurons. Inflammatory cytokines and the vagal system in turn can modulate the activity of the CNS and ENS.Neuro/immune-active substances derived from the intestinal lumen can penetrate the gut mucosa, be transported by blood, cross the blood-brain-barrier (BBB) and affect the CNS. Gut microbiota can influence CNS function through their ability to synthesize or mimic a range of host-signaling neuroactive molecules, such as acetylcholine (Ach), catecholamines, gamma-aminobutyric acid (GABA), histamine, melatonin and 5-hydroxytryptamine (5-HT, serotonin). 5-HT is crucial in the regulation of of peristalsis or modulation of sensation.

Parkinson's disease (PD) is a multicentric neurodegenerative disorder characterized by the accumulation and aggregation of alfa-synuclein (α-syn) in the substantia nigra in the central nervous system (CNS) and in other neural structures. The classical motor symptoms like bradykinesia, resting tremor, rigidity and late postural instability result from the death of dopamine-generating cells in the substantia nigra. There is also a wide spectrum of non-motor manifestations involving for example olfactory (loss of smell), gastrointestinal (GI), cardiovascular and urogenital systems. It has become evident that the different levels of the brain-gut axis including the autonomic nervous system (ANS) and the enteric nervous system (ENS) may be affected in PD. Recently, it has been also recognized that the brain-gut axis interactions may be essentially influenced by the gut microbiota. On the one hand, dysregulation of the brain-gut-microbiota axis in PD may result in GI dysfunction, which is present in over 80% of PD subjects . On the other hand, this dysregulation may also significantly contribute to the pathogenesis of PD itself, supporting the hypothesis that the pathological process is spread from the gut to the brain .

GUT MICROBIOTA AND PARKINSON'S DISEASE

Over the past decade, experimental data has suggested a complex and bidirectional interaction between the gastrointestinal (GI) tract and the central nervous system (CNS), the so-called "Gut- Brain axis." . Changes in the gut microbiota composition may cause alterations in the gut barrier function and intestinal permeability, affecting not only GI epithelial cells and immune system, but also the ENS including both neurons and glial cells . The bidirectional brain-gut-microbiota axis interactions modulate pro- and anti-inflammatory responses. It has been suggested that the gut microbiota changes associated with intestinal inflammation may contribute to the initiation of α-syn misfolding. There is a growing number of evidence confirming that the gut microbiota alterations precede or occur during the course of PD. However, the causal relationship between the microbiota changes and the pathogenesis of PD remains unclear.

The interesting concept of molecular mimicry involving the microbiota in neurodegeneration has been also proposed. Indeed, Friedland suggested that bacterial proteins may elicit cross-seeded misfolding, inflammation and oxidative stress, and cellular toxicity in neurodegeneration, initiating or otherwise influencing the development of PD, Alzheimer's disease and other related disorders. Pathways of molecular mimicry processes induced by bacterial amyloid may involve TLR2/1, C14, and NFκB among others. Priming of the innate immune system by the microbiota (residing in the gut and oral/nasal cavities) may enhance the inflammatory response to cerebral amyloids such as α-syn. Trudler et al postulated that cerebral amyloid may mimic viral or bacterial infection resulting in glial cell activation through TLRs. Specifically, it has been documented that neuroinflammation in PD is associated with upregulation of TLR2 signaling and activation of microglia. TLR2, playing an important role in the regulation of intestinal barrier integrity, has been also found to activate microglial cells in the CNS. It has been suggested that the peripheral immune response characterized by the presence of pro-inflammatory cytokines such as TNF-α, IL-1β and IL-8 in the serum induces a disruption of the blood-brain barrier and promotes microglia-mediated inflammation and neurotoxicity. In a germ-free animal model, it has been found that the gut microbiota influences the blood-brain barrier permeability associated with reduced expression of the tight junction proteins in a homological way as it affects the intestinal epithelial barrier. Very recently, Sui et al proved that a bidirectional transport of α-syn into and out of the brain by the blood-brain barrier is possible and suggested that LPS-induced inflammation could increase α-syn uptake by the brain by disrupting the blood-brain barrier.

In an animal model of PD, peripherally-induced inflammation was shown to induce the microglial complement pathway to damage dopaminergic neurons. Several studies have demonstrated that pro-inflammatory factors associated with chronic GI diseases induce brain inflammation and the death of dopaminergic neurons and could eventually be responsible for parkinsonism.

Importantly, some genetic risk factors may play a crucial role in the interactions between the brain-gut-microbiota axis with respect to gut inflammation. It has been also shown that the methylation status in the SNCA promoter region may affect α-syn expression and the risk for PD. Therefore, a potential role of the gut microbiota as an epigenetic factor influencing DNA methylation may be speculated. Moreover, genetic variant of the component of innate immune system - TREM2 (Triggering Receptor Expressed on Myeloid cells) has been reported to be associated with a higher risk for PD. The ε4 allele of apolipoprotein E (ApoE) has been shown to increase the risk for dementia in synucleinopathies such as PD. Potentially, ApoE genotype, by influencing bile acid secretion, could affect the composition of the gut microbiota to favor the development of organisms triggering misfolding. Moreover, three single nucleotide polymorphisms in CARD15 gene, known to be associated with Crohn's disease, have been also shown to be over-expressed in PD patients, supporting the observation that GI inflammation contributes to the pathogenesis of PD.

ELIGIBILITY:
Inclusion Criteria:

* (50) patients diagnosed with Parkinson's Disease .
* (50) Control group free from Disease .

Exclusion Criteria:

* prior surgeries.
* any patients or controls currently taking antibiotics or probiotic supplements.
* having a known history of disease with an disease such, autoimmune disorders , cardiac patients
* history of stroke ,rheumatoid arthritis, type-1-diabetes, and IBD .

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Unified Parkinson's Disease Rating Scale (UPDRS) and the modified Hoehn & Yahr Scale (H&Y). Non-Motor Symptoms Scale (NMSS).
  Demographic and clinical data (Age, sex, age of onset, severity of disease, clinical symptoms and signs, Types of treatment, duration of treatment, number of attacks)
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-01-01 (Estimated); Primary Completion 2020-01-01 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Effect of gut microbiota on pathogenesis of Parkinson's diseases | 1 year
  the QIAamp DNA Stool mini kit to extract total bactria DNA Some genetic risk factors may play a crucial role in the interactions between the brain-gut-microbiota axis with respect to gut inflammation. It has been also shown that the methylation status in the SNCA promoter region may affect α-syn expression and the risk for PD

IPD SHARING:
Plan to Share IPD: Undecided